CLINICAL TRIAL: NCT06351566
Title: Effects of Vitamin D3 and Prebiotics Supplementation on Cardiovascular Risk Factors in Patients With Type 2 Diabetes: A Randomized Double-Blind Controlled Trial
Brief Title: Effects of Vitamin D3 and Prebiotics Supplementation on Cardiovascular Risk Factors in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, An Pan, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VD3, Prebiotics in Diabetes
Record Dates: First submitted 2024-03-08; First posted 2024-04-08 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vitamin D; Prebiotics; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Blood Glucose; Lipids
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Cholecalciferol; Prebiotics; Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vitamin D3 + Prebiotics (Active Comparator)
  Interventions: Drug: Vitamin D3; Dietary Supplement: Prebiotics
- Vitamin D3 + Prebiotics placebo (Active Comparator)
  Interventions: Drug: Vitamin D3; Dietary Supplement: Prebiotics placebo
- Prebiotics +Vitamin D3 placebo (Active Comparator)
  Interventions: Dietary Supplement: Prebiotics; Dietary Supplement: Vitamin D3 placebo
- Vitamin D3 placebo + Prebiotics placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Prebiotics placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 (cholecalciferol), 1600 IU per day.
  Other Names: Cholecalciferol
  Arms: Vitamin D3 + Prebiotics; Vitamin D3 + Prebiotics placebo
Dietary Supplement: Prebiotics — Prebiotics (inulin), 10g per day.
  Other Names: Inulin
  Arms: Prebiotics +Vitamin D3 placebo; Vitamin D3 + Prebiotics
Dietary Supplement: Vitamin D3 placebo — Vitamin D3 placebo
  Arms: Prebiotics +Vitamin D3 placebo; Vitamin D3 placebo + Prebiotics placebo
Dietary Supplement: Prebiotics placebo — Prebiotics placebo, 10g per day.
  Arms: Vitamin D3 + Prebiotics placebo; Vitamin D3 placebo + Prebiotics placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled, 6-month supplementation study in individuals with type 2 diabetes is to investigate whether taking daily dietary supplements of vitamin D3 (1600 IU) or prebiotics (inulin, 10 gram) has beneficial effects on cardiovascular disease risk factors.

DETAILED DESCRIPTION:
The goal of this randomized, double-blind, placebo-controlled trial, with a two-by-two factorial design in individuals with type 2 diabetes (T2D) is to investigate whether taking daily dietary supplements of vitamin D3 (1600 IU) or prebiotics (inulin, 10 gram) has beneficial effects on cardiovascular disease (CVD) risk factors.

About 200 subjects with T2D will be included in this study. All participants will provide written informed consent before randomization. Eligible participants must have no history of cancer, macrovascular or microvascular complications at trial entry, and they are required to agree to limited use of vitamin D, prebiotics, probiotics, or synbiotic supplementations, as well as to convenient access to study centers. Safety exclusions include renal failure or dialysis, cirrhosis, history of hypercalcemia, or other conditions that would preclude participation.

Eligible participants will be assigned by chance to one of four groups: (1) daily vitamin D3 (1600 IU) and prebiotics (10 grams); (2) daily vitamin D3 (1600 IU) and prebiotics placebo (10 grams); (3) daily vitamin D3 placebo and prebiotics (10 grams); or (4) daily vitamin D3 placebo (1600 IU) and prebiotics placebo (10 grams). Randomization will be computer-generated within sex and age groups.

During the run-in period, baseline questionnaires will be designed to collect data on sociodemographic factors, lifestyle habits, health status, and medical conditions, and participants will undergo physical measurements at baseline. Blood, urine, and faeces samples will also be obtained at study centers.

Participants in all groups will be required to take two capsules each day, containing either vitamin D3 or vitamin D3 placebo, as well as a strip of prebiotics powder (10 g per strip, brew with warm water) or prebiotics placebo. Participants will receive their capsules and powder at study centers each month.

Participants will complete follow-up questionnaires, including information on adherence to trial regimens, outside use of supplementations, development of major illnesses, and potential side effects of the trial agents, at 3 months and 6 months after randomization. Physical measurements and collection of biological samples will be conducted at study centers 6 months after randomization.

The primary outcomes, including glycated hemoglobin (HbA1c) and blood lipids (such as total cholesterol, triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol), will be measured using blood samples. The data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes (meeting any of the following criteria):

   Physician-diagnosed type 2 diabetes, use of oral hypoglycemic medication or insulin, fasting blood glucose ≥ 7.0 mmol/L, HbA1c ≥ 6.5% (48 nmol/L), 2-hour plasma glucose (2hPG) ≥ 11.1 mmol/L.
2. Men aged 35-70 years or women aged 35-70 years.
3. Convenient access to study centers.
4. Written informed consent obtained before any trial-related activities.

Exclusion Criteria:

1. History of macrovascular diseases (including Coronary heart disease, myocardial infarction, heart failure, stroke, transient ischemic attack, peripheral vascular disease, post coronary artery bypass surgery).
2. History of diabetic microvascular complications (including diabetic nephropathy, diabetic retinopathy, or diabetic neuropathy).
3. History of other cardiovascular diseases (including aortic stenosis, transient ischemic attack, angina pectoris, cardiac arrest, complex ventricular arrhythmias, or surgery of cardiovascular diseases).
4. History of cancer, excluding non-melanoma skin cancer or cancers with a good prognosis (such as stage 1 cervical cancer).
5. Severe liver disease (such as cirrhosis), severe kidney disease (such as renal failure or requiring dialysis), or severe gastrointestinal disease (such as a history of bowel obstruction).
6. Kidney stones, hypercalcemia, parathyroid hormone abnormality.
7. Sarcoidosis or other granulomatous diseases, such as active chronic pulmonary tuberculosis or Wegener's granulomatosis.
8. Any mental disorders, such as schizophrenia, other mental disorders, or bipolar disorder.
9. Individuals with infectious diseases such as HIV/AIDS, viral hepatitis.
10. Individuals requiring long-term hospitalization or those with other serious illnesses requiring immediate hospital treatment.
11. In the past 3 months, those who have taken any vitamin D supplements exceeding 400 IU/day, calcium supplements exceeding 600 mg/day, prebiotics exceeding 2 g/day, or probiotics exceeding 10^8 colony forming units/day.
12. History of allergy or intolerance to vitamin D, prebiotics, or starch.
13. Individuals with unhealthy habits: heavy alcohol consumption (>80 grams/day for males, >40 grams/day for females) or smoking (>40 cigarettes/day).
14. Individuals with cognitive impairment, inability to communicate properly, inability to take care of themselves, or those with mobility issues.
15. Those having participated in other clinical trials or studies in the past 3 months.
16. Those who are intent to become pregnant within the next two years, are currently pregnant, or breastfeeding.
17. Individuals with abnormal laboratory tests and clinical manifestations who are judged by the researcher to be unsuitable for participation.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 6 months
  Concentration of HbA1c, measured in the percentage of hemoglobin
Concentration of blood lipids | 6 months
  Concentration of blood lipids (total cholesterol, triglycerides, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol), measured in mmol/L
Metagenomic analysis of the gut microbiota | 6 months
  The diversity of the gut microbiota will be assessed by high-quality whole-metagenomic sequencing

SECONDARY OUTCOMES:
Concentration of fasting glucose | 6 months
  Concentration of fasting glucose, measured in mmol/L
Concentration of fasting insulin | 6 months
  Concentration of fasting insulin, measured in milli-International unit/L
Systolic and diastolic blood pressure | 6 months
  The level of systolic blood pressure and diastolic blood pressure, measured in mmHg
Estimated glomerular filtration rate (eGFR) | 6 months
  Calculating the level of eGFR using Chronic Kidney Disease Epidemiology Collaboration equation
Concentration of C-reactive protein (CRP) | 6 months
  Concentration of CRP, measured in mg/dL
Concentration of procalcitonin | 6 months
  Concentration of procalcitonin, measured in pg/mL
Concentration of interleukin-6 (IL-6) | 6 months
  Concentration of IL-6, measured in pg/mL
Concentration of serum 25(OH)D | 6 months
  Concentration of serum 25(OH)D concentrations, measured in nmol/L
Body weight | 6 months
  Weight in kilograms
Waist circumference | 6 months
  Waist circumference in centimeters
Hip circumference | 6 months
  Hip circumference in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Gang Liu, PHD, Principal Investigator — School of Public Health, Tongji Medical College, Huazhong University of Science and Technology; An Pan, PHD, Principal Investigator — School of Public Health, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Bao'an Center Hosipital of Shenzhen, Shenzhen, Guangdong
  - School of Public Health, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No